CLINICAL TRIAL: NCT07044778
Title: Prevalence And Risk Factor Of Overactive Bladder Syndrome Among Egyptian Medical Students And Their Impact On Health-Related Quality Of Life, Cross-Sectional Study
Brief Title: Prevalence And Risk Factors of Overactive Bladder Syndrome Among Egyptian Medical Students, and Their Impact On Health-Related Quality Of Life
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Other Study IDs: ZU-IRB # 1328 /18-May-2025
Record Dates: First submitted 2025-05-24; First posted 2025-07-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-05

CONDITIONS: Overactive Bladder Syndrome
Keywords: overactive bladder; Prevalence; medical students; quality of life
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — An online Questionnaire designed by Google Forms will be shared on social media for medical students in Egypt to fill

SUMMARY:
Overactive bladder (OAB) is defined as sudden, urgent desire to urinate (urgency) accompanied by frequency and nocturia, with or without urgent urinary incontinence in the absence of urinary tract infection (UTI). This condition can significantly decrease the quality of life of these patients, as it can humiliate their actions, affect their relationships with others, and it can also affect their productivity. Due to all these effects, several studies have linked the increase in overactive bladder symptoms with an increase in anxiety and depression rates. A recent cross-sectional study in the UK and Sweden, called EpiLUTS, included 10,000 participants. the investigators found a statistically significant increase in anxiety and depression rates among both men and women in both the UK and Sweden, with a slight increase in men than women On the other hand, there are several risk factors such as overweight, smoking, diabetes, and hypertension. In a previous cross-sectional study in Jordan, the investigators found a correlation between an increase in risk factors such as age group, history of trauma, stressful life, and medication, and overactive bladder symptoms among medical students.

Several studies have assessed the prevalence of overactive bladder among different population age groups, ethnicities, or genders with varying results. It was rated to be 11.8% in a multicenter cross-sectional study including several countries in Canada and Europe (Germany, Italy, Sweden, and the UK), while in the USA it was estimated to be 16%. All these studies were conducted on the general population; however, in China, it was about 6% among university students.

In the Arab world, several cross-sectional studies have also assessed the prevalence of overactive bladder, including students, and its effect on the quality of life. Hajjar 2022 assessed its prevalence among Lebanese female nulliparae university students. They showed that nocturia and frequency were the most common symptoms that bothered students. the investigators also found a statistical correlation between smoking, drinking coffee, or tea, and increased symptoms. Also, drinking soft drinks was associated with an increase in urinary leakage. Additionally, Abuorouq 2024 and Shawahna 2021 conducted Cross-sectional studies were conducted on medical students in Jordan and Palestine, respectively. They reported a prevalence of 44.5% and 54.1%, respectively. Shawahna 2021 reported a statistically significant correlation between gender or stressful life and a decrease in quality of life.

Rational In Egypt, the prevalence of overactive bladder is underestimated. A single previous multinational cross-sectional study across several Arab countries, including Egypt, was conducted. was conducted in Egypt, Algeria, Jordan, and Lebanon among women. the investigators reported a prevalence of 57.5% among Egyptian women.

Since this study, no study has been conducted to further assess its prevalence in different age or gender groups in Egypt. Taking into consideration the stressful life of medical students in Egypt, and several life risk factors they face, the investigators will conduct this cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* Medical student studying human medicine in Egypt
* Their age ranges from 18 to 27 years old
* Egyptian person

Exclusion Criteria:

* Incomplete data
* Wrong data in the questionnaire
* Students refuse to participate

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Egyptian medical students who have access to social media
Sampling Method: Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Overactive Bladder Syndrome prevalence | through study completion, an average of 1 month
  We will use OAB-q SF for diagnosing symptoms bother. It is a 6-item questionnaire to diagnose symptoms bother; each question has 6 Likert scale answers. A score of 1 to 6 for each question will form a scale of 6 to 36. An increase in score indicates an increase in symptoms bother

SECONDARY OUTCOMES:
Quality of life affected by OAB | through study completion, an average of 1 month
  Using the second part of the OAB-q SF (HRQL). This is a 13 Likert scale questionnaire. each question has 6 answers to assess its quality of life. A score range from 13 to 78, with a decrease indicating a decrease in the quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- All Egypt, Zagazig, Egypt

REFERENCES:
- [Result] Coyne KS, Payne C, Bhattacharyya SK, Revicki DA, Thompson C, Corey R, Hunt TL. The impact of urinary urgency and frequency on health-related quality of life in overactive bladder: results from a national community survey. Value Health. 2004 Jul-Aug;7(4):455-63. doi: 10.1111/j.1524-4733.2004.74008.x. PMID 15449637
- [Result] Abuorouq S, Al-Zubi M, Al-Ali AM, Aloqaily LH, Talafha MA, Migdadi AM, Serhan HA. The prevalence of probable overactive bladder and associated risk factors among medical students in Jordan: a cross-sectional study. BMC Urol. 2024 Jan 3;24(1):7. doi: 10.1186/s12894-023-01394-4. PMID 38172746

DOCUMENTS (1):
  • Study Protocol (2025-05-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT07044778/Prot_000.pdf